CLINICAL TRIAL: NCT07072611
Title: A Double-Blind, Placebo-Controlled Phase I Clinical Trial to Evaluate Safety, Tolerability, and Pharmacokinetics of SOF-SKN in Healthy Participants
Brief Title: Clinical Trial to Evaluate Safety, Tolerability, and Pharmacokinetics of SOF-SKN in Healthy Participants
Acronym: HERACLES
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Noxopharm Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PHA-001
Record Dates: First submitted 2025-06-16; First posted 2025-07-18 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-06

CONDITIONS: Cutaneous Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Cutaneous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Cohort 1 (Active Comparator): Single application of 2 g SOF-SKN cream 2.5 mg/g (0.25% w/w) applied topically to 10 × 30 cm area on the left or right side of the participant's back. In addition, a single 2 g application of placebo cream, to serve as an intra-participant control, will be applied to a 10 × 30 cm area on the alternate side of the participant's back.
  Interventions: Drug: SOF-SKN 0.25%; Drug: Placebo
- Cohort 2 (Active Comparator): Single application of 2 g SOF-SKN cream 5 mg/g (0.5% w/w) applied topically to 10 × 30 cm area on the left or right side of the participant's back. In addition, a single 2 g application of placebo cream, to serve as an intra-participant control, will be applied to a 10 × 30 cm area on the alternate side of the participant's back.
  Interventions: Drug: SOF-SKN 0.5%; Drug: Placebo
- Cohort 3 (Active Comparator): Single application of 2 g SOF-SKN cream 10 mg/g (1% w/w) applied topically to 10 × 30 cm area on the left or right side of the participant's back. In addition, a single 2 g application of placebo cream, to serve as an intra-participant control, will be applied to a 10 × 30 cm area on the alternate side of the participant's back.
  Interventions: Drug: SOF-SKN 1%; Drug: Placebo
- Cohort 4 (Active Comparator): Single application of 2 g SOF-SKN cream 20 mg/g (2% w/w) applied topically to 10 × 30 cm area on the left or right side of the participant's back. In addition, a single 2 g application of placebo cream, to serve as an intra-participant control, will be applied to a 10 × 30 cm area on the alternate side of the participant's back.
  Interventions: Drug: SOF-SKN 2%; Drug: Placebo
- Cohort 5 (Active Comparator): Multiple applications of 2 g SOF-SKN cream 2.5 mg/g (0.25% w/w) once a day over 14 days applied topically to 10 × 30 cm area on the left or right side of the participant's back. In addition, a single 2 g application of placebo cream, to serve as an intra-participant control, will be applied to a 10 × 30 cm area on the alternate side of the participant's back.
  Interventions: Drug: SOF-SKN 0.25%; Drug: Placebo
- Cohort 6 (Active Comparator): Multiple applications of 2 g SOF-SKN cream 5 mg/g (0.5% w/w) once a day over 14 days applied topically to 10 × 30 cm area on the left or right side of the participant's back. In addition, a single 2 g application of placebo cream, to serve as an intra-participant control, will be applied to a 10 × 30 cm area on the alternate side of the participant's back.
  Interventions: Drug: SOF-SKN 0.5%; Drug: Placebo
- Cohort 7 (Active Comparator): Multiple applications of 2 g SOF-SKN cream 10 mg/g (1% w/w) once a day over 14 days applied topically to 10 × 30 cm area on the left or right side of the participant's back. In addition, a single 2 g application of placebo cream, to serve as an intra-participant control, will be applied to a 10 × 30 cm area on the alternate side of the participant's back.
  Interventions: Drug: SOF-SKN 1%; Drug: Placebo
- Cohort 8 (Active Comparator): Multiple applications of 2 g SOF-SKN cream 20 mg/g (2% w/w) once a day over 14 days applied topically to 10 × 30 cm area on the left or right side of the participant's back. In addition, a single 2 g application of placebo cream, to serve as an intra-participant control, will be applied to a 10 × 30 cm area on the alternate side of the participant's back.
  Interventions: Drug: SOF-SKN 2%; Drug: Placebo

INTERVENTIONS:
Drug: SOF-SKN 0.25% — cream for topical application
  Arms: Cohort 1; Cohort 5
Drug: SOF-SKN 0.5% — cream for topical application
  Arms: Cohort 2; Cohort 6
Drug: SOF-SKN 1% — cream for topical application
  Arms: Cohort 3; Cohort 7
Drug: SOF-SKN 2% — cream for topical application
  Arms: Cohort 4; Cohort 8
Drug: Placebo — cream for topical application

SUMMARY:
The goal of this study is to investigate the safety and tolerability of the topical application of SOF-SKN in healthy volunteers. The study will be divided into part 1 and part 2.

Part 1, is a single ascending dose (SAD) design, while Part 2 is a multiple ascending dose (MAD) design.

DETAILED DESCRIPTION:
The study will contain four, single ascending dose-escalation cohorts and four multiple dose-escalation cohorts allowing an exploration of different doses of SOF-SKN with safety monitoring to ensure the safety of the participants.

A maximum of thirty-two (32) participants will be enrolled overall, with a maximum of sixteen (16) participants enrolled into each part of the study.

There is to be a 28-day Screening period (Day -28 to -1) for both Part 1 and 2 of the study.

Both SAD and MAD will include four treatment cohorts (0.25%, 0.5%, 1% and 2%) of SOF-SKN.

Participants enrolled Part 1 (SAD) will receive a single dose of 2 g Soft-SKN cream while the participants enrolled in Part 2 (MAD) will receive daily applications of 2 g SOF-SKN cream for 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers 18 to 64 years.
* Participants with Fitzpatrick skin type I to IV.
* Participants must have a back surface area of at least 24 × 30 cm to accommodate two - 10 × 30 cm application areas with a 4 cm separation between them.
* No Allergies.
* Contraception.
* Must be willing to abstain from the use of moisturizers and other topical applications on the back 24 hours prior and for the duration of the study.

Exclusion Criteria:

* Allergic constitution.
* Within 72 hours of the start of study treatment, the use of antihistamines or use of topical drugs at the application site.
* Hair removing interventions including laser treatment, shaving and waxing in the target area within 1 week before Screening.
* Hypertrichosis on the back; no tattoos that cover greater than 30% of the back surface area.
* Presence of an inflammatory dermatosis (including, but not limited to, atopic dermatitis, eczema, psoriasis, extensive acne), and/or suntan/burn that could interfere with the test field evaluation.
* Non-inflammatory skin lesions and changes (including, but not limited to, hyperpigmentation, multiple naevi, tattoos, blemishes, birthmarks, abrasions, ulcers, eschar, and/or scabs) present in the target area on the back that could interfere with the test field evaluation.
* Any history of or presence of in situ melanoma and non-melanoma skin cancer within the last 3 years.
* Any other skin disease or other visible skin condition noted on physical examination which in the Investigator's opinion might interfere with the evaluation of the test field reaction.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of Target Toxicities after a single treatment | 4 days -3 days after last application of topical treatment
  Part 1: Percentage of Target Toxicities after a single application of study treatment
Percentage of Target Toxicities after two-week treatment | 17 days - 3 days after last dose of treatment
  Part 2: Percentage of Target Toxicities following two weeks of daily application of study treatment
Percentage of Adverse events (AEs) after a single treatment | 4 days -3 days after last application of topical treatment
  Part 1: Percentage of AEs after a single application of study treatment
Percentage of Adverse events (AEs) after two-week treatment | 17 days - 3 days after last dose of treatment
  Part 2: Percentage of AEs following two weeks of daily application of study
Percentage of Serious Adverse events (SAEs) after a single treatment | 4 days -3 days after last application of topical treatment
  Part 1: Percentage of SAEs after a single application of study treatment
Percentage of serious Adverse events (SAEs) after two-week treatment | 17 days - 3 days after last dose of treatment
  Part 2: Percentage of SAEs following two weeks of daily application of study treatment.

SECONDARY OUTCOMES:
Maximum Tolerated Dose (MTD) of a single application of SOF-SKN | 4 days -3 days after last application of topical treatment
  To determine the MTD of a single application of SOF-SKN cream.
Maximum Tolerated Dose (MTD) for multiple applications of SOF-SKN | 17 days - 3 days after last dose of treatment
  To determine the MTD of multiple applications following two weeks of daily application of study treatment with SOF-SKN cream.
Maximum concentration (Cmax) of a single application of SOF-SKN | 7 timepoints from baseline to 24 hours (baseline, 30 mins, 1, 2, 4, 6 and 24 hours)
  PK parameters will be calculated to determine the degree of systemic exposure. The Maximum concentration (Cmax) will be calculated, if possible, as minimal systemic exposure is expected.
Time to reach Cmax (tmax) of a single application of SOF-SKN | 7 timepoints from baseline to 24 hours (baseline, 30 mins, 1, 2, 4, 6 and 24 hours)
  PK parameters will be calculated to determine the degree of systemic exposure. Time to reach Cmax (tmax), if possible, as minimal systemic exposure is expected.
Area Under the Concentration-Time Curve (AUC) of a single application of SOF-SKN | 7 timepoints from baseline to 24 hours (baseline, 30 mins, 1, 2, 4, 6 and 24 hours)
  PK parameters will be calculated to determine the degree of systemic exposure. The Area Under the Concentration-Time Curve (AUC) will be calculated from Time Zero to the Last Measurable Plasma Concentration (AUC0-last), if possible, as minimal systemic exposure is expected.
AUC Extrapolated to Infinity (AUC0-inf) of a single application of SOF-SKN | 7 timepoints from baseline to 24 hours (baseline, 30 mins, 1, 2, 4, 6 and 24 hours)
  PK parameters will be calculated to determine the degree of systemic exposure. The AUC Extrapolated to Infinity (AUC0-inf) will be calculated, if possible, as minimal systemic exposure is expected.
Half-life (t1/2) of a single application of SOF-SKN | 7 timepoints from baseline to 24 hours (baseline, 30 mins, 1, 2, 4, 6 and 24 hours)
  PK parameters will be calculated to determine the degree of systemic exposure. The Half-life (t1/2) will be calculated, if possible, as minimal systemic exposure is expected.
Maximum concentration (Cmax) for multiple applications of SOF-SKN | 7 timepoints from baseline to day 17 (baseline, Day 1, Day 2, Day 4, Day 7, Day 10, Day 14 and Day 17)
  PK parameters will be calculated to determine the degree of systemic exposure The Maximum concentration (Cmax) will be calculated, if possible, as minimal systemic exposure is expected.
Time to reach Cmax (tmax) for multiple applications of SOF-SKN | 7 timepoints from baseline to day 17 (baseline, Day 1, Day 2, Day 4, Day 7, Day 10, Day 14 and Day 17)
  PK parameters will be calculated to determine the degree of systemic exposure The Time to reach Cmax (tmax) will be calculated, if possible, as minimal systemic exposure is expected.
Area Under the Concentration-Time Curve (AUC) for multiple applications of SOF-SKN | 7 timepoints from baseline to day 17 (baseline, Day 1, Day 2, Day 4, Day 7, Day 10, Day 14 and Day 17)
  PK parameters will be calculated to determine the degree of systemic exposure The Area Under the Concentration-Time Curve (AUC) Calculated from Time Zero to the Last Measurable Plasma Concentration (AUC0-last) will be calculated, if possible, as minimal systemic exposure is expected.
AUC Extrapolated to Infinity (AUC0-inf) for multiple applications of SOF-SKN | 7 timepoints from baseline to day 17 (baseline, Day 1, Day 2, Day 4, Day 7, Day 10, Day 14 and Day 17)
  PK parameters will be calculated to determine the degree of systemic exposure The AUC Extrapolated to Infinity (AUC0-inf) will be calculated, if possible, as minimal systemic exposure is expected.
Half-life (t1/2) for multiple applications of SOF-SKN | 7 timepoints from baseline to day 17 (baseline, Day 1, Day 2, Day 4, Day 7, Day 10, Day 14 and Day 17)
  PK parameters will be calculated to determine the degree of systemic exposure The Half-life (t1/2) will be calculated, if possible, as minimal systemic exposure is expected.
Drug Accumulation Ratio (Rac) for multiple applications of SOF-SKN | 7 timepoints from baseline to day 17 (baseline, Day 1, Day 2, Day 4, Day 7, Day 10, Day 14 and Day 17)
  PK parameters will be calculated to determine the degree of systemic exposure The Drug Accumulation Ratio (Rac) will be calculated, if possible, as minimal systemic exposure is expected.

CONTACTS AND LOCATIONS:
Locations (1):
- Doherty Clinical Trials, Melbourne, Victoria, Australia